CLINICAL TRIAL: NCT07307924
Title: The Effect of Motivational Interviewing on Knowledge, Self-Efficacy, and Treatment Adherence in Patients With Primary Hypertension Living in Semi-Rural Areas: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing on Knowledge, Self-Efficacy, and Treatment Adherence in Patients With Primary Hypertension Living in Semi-Rural Areas
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Şenay ÖZER, Lecturer and PhD Candidate, Eskisehir Osmangazi University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-190026
Record Dates: First submitted 2025-11-17; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Individuals (Controls); PRIMARY HYPERTENSION PATIENT
Keywords: Primary Hypertension; Motivational Interviewing; Knowledge Level; Self-Efficacy Level; Adherence to Treatment; Randomized Controlled Trial
MeSH Terms: conditions — Essential Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: A Health Belief Model-based motivational interviewing (MI) program will be implemented for participants assigned to the intervention group. Previous studies examining MI-guided nursing interventions in individuals with hypertension have predominantly adopted randomized controlled trial (RCT) designs and have emphasized individualized, patient-centered approaches. Although the duration, structure, and delivery methods of MI-based interventions vary across studies, these programs are generally designed as multifaceted and structured strategies that promote treatment adherence and support lifestyle modification.
  In alignment with this evidence, the MI program developed for the present study will consist of four sessions delivered over a maximum period of eight weeks. Sessions will take place biweekly and are planned to last between 30 and 45 minutes each.
Who Masked: Outcomes Assessor
Masking Description: In this study, participants were blinded to their assignment to the intervention or control group, thereby ensuring a single-blind design. As the research was conducted as part of a doctoral dissertation, the investigator personally carried out both the data collection procedures and the delivery of the intervention. For this reason, blinding during the implementation phase was not feasible. Nevertheless, to minimize potential bias, data entry and all statistical analyses were performed independently and in a blinded manner by a statistician who was not involved in any other stage of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Motivational interviewing) (Active Comparator): A four-session intervention based on the Health Belief Model (HBM) and delivered through motivational interviewing (MI) will be provided to the intervention group. The program aims to enhance risk perception, improve treatment adherence, strengthen self-efficacy, and support lifestyle change. The first session reviews hypertension and its risks to increase perceived susceptibility and severity. The second highlights treatment benefits, medication adherence, and key lifestyle modifications. The third focuses on building self-efficacy through personalized goals and an action plan supported by tools such as blood pressure diaries. The final session reinforces motivation, evaluates progress, and introduces relapse-prevention strategies. Sessions are held biweekly, last 30-45 minutes, and are supported by structured educational materials.
  Interventions: Behavioral: Motivasyonel görüşme
- Control Arm (No Intervention): In the control group, no educational content, counseling, or motivational interviewing was provided; participants continued with standard routine care only. Baseline, mid-intervention, and post-intervention assessments were conducted concurrently with the intervention group and included the administration of a sociodemographic information form, the Hypertension Knowledge Level Scale, the Hill-Bone Medication Adherence Scale, and the Hypertension Self-Efficacy Scale, along with standardized measurements of systolic and diastolic blood pressure. The control group served as a non-intervention comparator, allowing the natural course of patient adherence and self-management to be observed. This design ensured that any differences observed between groups could be attributed to the structured intervention rather than external influences.

INTERVENTIONS:
Behavioral: Motivasyonel görüşme — Hipertansiyon hastalarında yaşam tarzı değişikliklerinin teşvik edilmesi, tedaviye uyumun artırılması ve öz yeterlilik düzeylerinin geliştirilmesine yönelik yapılandırılmış müdahale programları, son yıllarda literatürde önemli yer edinmiştir.
  Sonuç olarak, MG tabanlı müdahaleler süre, içerik ve uygulama araçları bakımından çeşitlilik gösterse de, katılımcıların tedaviye uyumunu ve yaşam tarzı değişikliklerini desteklemek üzere çok yönlü ve yapılandırılmış programlar olarak öne çıkmaktadır. Bu bağlamda, çalışmamızda SİM temelli MG programının maksimum 8 hafta süresince, iki haftada bir olacak şekilde 4 oturumdan oluşacak ve her oturumun 30 ila 45 dakika arasında değişen sürelerde gerçekleştirilmesi planlanmaktadır. Eğitim içeriği, katılımcıların bilişsel düzeyleri, sağlık algıları ve davranış değişimine yönelik motivasyon düzeyleri dikkate alınarak yapılandırılmıştır.
  Arms: Intervention Arm (Motivational interviewing)

SUMMARY:
This study is a single-center, single-blind, parallel-group randomized controlled trial designed to examine the impact of a Health Belief Model (HBM)-based motivational interviewing (MI) intervention on knowledge level, self-efficacy, and treatment adherence among primary hypertension patients living in a semi-rural region. Hypertension, despite its typically asymptomatic course, is a prevalent chronic condition that contributes significantly to cardiovascular morbidity and mortality. Poor adherence to treatment and insufficient disease-related knowledge remain major barriers to achieving optimal blood pressure control. Self-efficacy is recognized as a crucial psychological determinant influencing lifestyle modification and medication adherence, and theoretical models-particularly the HBM-provide a structured framework for understanding individuals' health perceptions and facilitating behavioral change.

Motivational interviewing, a patient-centered counseling method aimed at strengthening intrinsic motivation, is thought to be particularly effective when combined with the HBM. The integration of these two approaches is expected to enhance individuals' readiness for change and promote active engagement in treatment. Existing evidence indicates that MI-based interventions can improve medication adherence, encourage lifestyle modifications, increase self-efficacy, and support better blood pressure control. These findings form the conceptual basis of the present study.

The trial was conducted between November 2025 and April 2026 at Hisarardı Family Health Center in Simav, Kütahya. The target population consisted of 140 individuals diagnosed with primary hypertension. Using G*Power with an effect size of 0.60, 80% power, and α=0.05, the required sample size was calculated as 50 participants per arm. Stratified randomization by sex and block randomization with blocks of four were employed.

The intervention group received a four-session MI program structured according to the HBM, consisting of the following components:

Enhancing risk perception and awareness of disease severity Highlighting treatment benefits and reducing perceived barriers Strengthening self-efficacy and developing a personalized action plan Strategies for maintaining behavioral change and identifying cues to action Each session lasted 30-45 minutes and was delivered biweekly. Participants in the control group did not receive any educational intervention and continued with routine clinical follow-up only.

Data were collected using the following instruments:

Hypertension Knowledge Level Scale Hill-Bone Medication Adherence Scale Hypertension Self-Efficacy Scale Systolic and diastolic blood pressure measurements Assessments were conducted at baseline (0 month), mid-intervention (3 months), and at the end of follow-up (6 months). Statistical analyses will be performed using SPSS 26.0, including paired and independent sample tests, correlation analyses, and effect size calculations.

Ethics approval, institutional permissions, and scale-use authorizations were obtained prior to data collection, and all procedures were carried out in accordance with the Declaration of Helsinki.

This study is expected to offer valuable insights into the applicability of theory-driven educational interventions in primary care settings, clarify the contribution of motivational interviewing to hypertension management, and inform national initiatives such as the Disease Management Platform (HYP).

DETAILED DESCRIPTION:
Hypertension is a chronic condition characterized by persistently elevated arterial blood pressure. It is clinically defined as a systolic blood pressure of ≥140 mmHg and/or diastolic pressure of ≥90 mmHg. The Turkish Society of Hypertension and Kidney Diseases (THBHD) emphasizes that hypertension often progresses silently without overt symptoms, yet over time it can lead to serious complications such as cardiovascular disease, stroke, renal failure, and other forms of target-organ damage.

Globally, hypertension is among the most prevalent chronic diseases and remains one of the leading contributors to cardiovascular morbidity and mortality. According to the World Health Organization, one in every three adults worldwide is living with hypertension. In Türkiye, the prevalence among adults aged 30-79 years is estimated at approximately 32%. Similarly, Şengül et al. reported a national prevalence of 30.3%.

Long-term hypertension management is closely linked to individuals' capacity to engage in lifestyle modifications, adhere to pharmacological treatment, and effectively self-manage their condition. However, numerous studies indicate that poor adherence to antihypertensive therapy and insufficient disease-related knowledge hinder optimal blood pressure control. These findings underscore the importance of understanding the beliefs and perceptions that shape individuals' health behaviors and developing structured educational models tailored to these determinants.

Self-efficacy, a key psychological construct in behavior change and chronic disease management, refers to an individual's belief in their ability to successfully perform a desired behavior. Evidence suggests that self-efficacy plays a central role in maintaining blood pressure control by enhancing medication adherence, reducing dietary sodium intake, supporting adherence to the DASH diet, promoting regular physical activity, and ensuring consistent blood pressure monitoring. Successful chronic disease management requires more than pharmacotherapy; individuals' disease perceptions, treatment attitudes, and health-related behaviors directly influence clinical outcomes.

Studies on chronic diseases such as hypertension demonstrate that individuals with strong self-efficacy are more committed to medication adherence, regular exercise, dietary adjustments, and self-monitoring behaviors. Accordingly, theoretical models that systematically explain health behaviors serve as valuable tools for guiding behavioral interventions. One such model, the Health Belief Model (HBM), conceptualizes individuals' perceptions of disease risk and the factors influencing engagement in health-promoting behaviors. The model comprises six constructs: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cues to action, and self-efficacy. Structured interventions based on these constructs have been shown to positively influence health behaviors and improve chronic disease outcomes, including in hypertension management.

Motivational interviewing (MI) is a complementary approach that strengthens the effectiveness of HBM-based interventions. MI is a collaborative, patient-centered counseling method that enhances intrinsic motivation for behavior change. Originally developed by Miller and Rollnick (1991) for substance use treatment, it is now widely employed in chronic disease management. MI helps individuals explore personal strengths, resolve ambivalence, and gain ownership of the change process, thereby reinforcing self-efficacy and supporting sustainable health behaviors.

Core principles of MI include demonstrating empathy, encouraging discrepancy between current behaviors and long-term goals, working constructively with resistance rather than confronting it, and enhancing self-efficacy. MI has been especially effective among individuals with low motivation, facilitating adoption and maintenance of health behaviors. In hypertension, MI has been shown to improve medication adherence, dietary compliance, exercise behaviors, and blood pressure monitoring.

When MI is integrated with the Health Belief Model, cognitive constructs such as perceived susceptibility and severity can be strengthened alongside self-efficacy, ultimately enhancing individuals' willingness to initiate and maintain behavioral change.

Primary care represents the foundational level at which preventive, continuous, and person-centered health services are delivered. For chronic conditions such as hypertension, implementing structured interventions that are responsive to individual belief systems and supportive of behavior change is essential. In this context, MI provides a patient-centered communication strategy that promotes treatment adherence, encourages active participation in disease management, and may help reduce the long-term burden on the healthcare system.

Recent studies indicate that MI interventions aligned with the Health Belief Model enhance patient awareness, support hypertension management, improve blood pressure control, strengthen self-efficacy, facilitate lifestyle behavior change, and significantly improve treatment adherence.

The primary aim of the present study is to evaluate the impact of motivational interviewing on knowledge level, self-efficacy, and treatment adherence among individuals diagnosed with primary hypertension living in a semi-rural area.

By integrating MI's motivational strategies with the HBM's focus on health perceptions, the study seeks to address both psychological and behavioral barriers to disease management and offer a theory-driven, practical solution to an important public health problem. It is anticipated that participants will achieve improved disease-related knowledge and awareness, enhanced adherence to treatment, and strengthened self-management abilities. These improvements are expected to promote sustainable lifestyle changes, better blood pressure control, a reduction in complication risk, and an overall improvement in quality of life.

The findings are expected to inform the national Disease Management Platform (HYP), support the feasibility of model-based educational programs in primary care, and contribute to evidence-based patient education practices that strengthen chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with primary hypertension,
* Being between 25 and 59 years of age,
* Having had a confirmed primary hypertension diagnosis for at least 12 months,
* Being literate and able to communicate in Turkish,
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Having cognitive impairment, dementia, or a severe psychiatric diagnosis,
* Having a diagnosis of secondary hypertension,
* Being pregnant or in the breastfeeding period,
* Having a physical disability or communication problem that would prevent active participation in the educational sessions.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In the study, to ensure an equal and homogeneous distribution of participants into the intervention and control groups, the 140 individuals in the sample were allocated using stratified randomization, based on baseline prognostic factors, particularly sex. Accordingly, the intervention group was composed of 50 participants-25 women and 25 men-and the control group was structured in the same manner, with 25 women and 25 men who shared similar baseline characteristics.
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
The knowledge levels of individuals in the intervention group demonstrate a significant increase after the training compared with those in the control group. | March 2026 (3 months later)
  The knowledge levels of individuals in the intervention group show a significant increase after the training compared with those in the control group.
The knowledge levels of individuals in the intervention group increase significantly after the training compared with those in the control group. | June 2026 (6 months after onset)
  The knowledge levels of individuals in the intervention group show a significantly greater increase after the training compared with those in the control group.

OTHER OUTCOMES:
The knowledge levels of individuals in the intervention group increase significantly after the training compared with those in the control group. | March 2026 (3 months later)
  The knowledge levels of individuals in the intervention group increase significantly after the training compared with those in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem ÖRSAL, PROF, Study Director — ESKİŞEHİR OSMANGAZİ UNIVERSITY INSTITUTE OF HEALTH SCIENCES DEPARTMENT OF NURSING
Locations (1):
- Hisarardı Family Health Center affiliated with the Simav District Health Directorate, Kütahya, Kütahya/ Simav, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Kasım 2025 - Aralık 2026

REFERENCES:
- See also: World Health Organization. (2023a). Global report on hypertension: The race against a silent killer. World Health Organization — https://iris.who.int/handle/10665/372896
- See also: World Health Organization (2023b). Hypertension — https://www.who.int/news-room/fact-sheets/detail/hypertension
- See also: World Health Organization. (2023c). Primary health care — https://www.who.int/health-topics/primary-health-care